CLINICAL TRIAL: NCT07119047
Title: Brazilian Adaptation of an Intervention Developed in Ireland to Promote Healthy Lifestyle Behaviors Post-stroke: Protocol for a Feasibility Study
Brief Title: Brazilian Adaptation of an Intervention Developed in Ireland to Promote Healthy Lifestyle Behaviors Post-stroke: a Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: FAPEMIG - Fundação de Amparo a Pesquisa do Estado de Minas Gerais (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenaçao de Aperfeiçoamento de Pessoal de Nível Superior (Unknown); Worldwide Universities Network (Unknown); Pró-reitoria de Pesquisa da Universidade Federal de Minas Gerais (Unknown)
Responsible Party: Principal Investigator, Christina Danielli Coelho de Morais Faria, Doctor, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 77083023.0.0000.5149
Record Dates: First submitted 2025-06-13; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Stroke; Healthy Lifestyle; Feasibility Study; Clinical Trial; Secondary Prevention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Brazilian adaptation of the Irish intervention "iHELP Stroke" (Experimental): The adaptation process of the Irish intervention "iHELP Stroke: Improving Health and Lifestyle Programme" for the Brazilian context followed the recommendations outlined in the ADAPT guidance (Moore et al., 2021). The adaptations proposed, discussed, and implemented aimed to tailor the intervention to Brazilian specificities, including geographic, cultural, economic, ethical, legal, political, organizational, service-related, and practice-related factors. Participants will undergo the Brazilian version of the adapted "iHELP Stroke" intervention over eight weeks. This includes one educational session (one hour), an initial individual session (one hour), and six group sessions (two hours each), totaling eight weeks of intervention.
  Interventions: Behavioral: A Brazilian adaptation of the Irish intervention "iHELP Stroke"

INTERVENTIONS:
Behavioral: A Brazilian adaptation of the Irish intervention "iHELP Stroke" — The intervention comprises a set of interactive experiential learning activities. A physiotherapist will serve as the coordinator, and other healthcare professionals will be invited to participate as guest speakers. The educational session aims to provide knowledge about stroke (what stroke and recurrent stroke are, their signs and symptoms, and lifestyle-related risk factors). The individual session aims: (1) to identify the current self-reported health status after stroke; (2) to recognize and raise awareness of risk factors associated with lifestyle-related behaviors, including the setting of behavior change goals, which are structured using the SMART Goals method; and (3) to identify the individual's preferences and ability to participate in the intervention program. Each group session comprises six components covered across the six sessions: education, goal setting, physical activity participation, emotional self-regulation, skill training, and peer learning.

SUMMARY:
Introduction: Low- and middle-income countries, such as Brazil, are most impacted by the high burden of recurrent stroke. These countries also lack structured interventions to promote the adoption of healthy lifestyle behaviors in the context of stroke secondary prevention. In contrast, high-income countries, such as Ireland, which invest more in research, have more advanced studies on this topic. However, before implementing interventions developed in countries like Ireland in middle-income countries like Brazil, it is necessary to adapt them to account for cultural and socioeconomic differences. Furthermore, once the adaptation is made, it is essential to investigate the feasibility of implementing the intervention in the new context.

Objective: To investigate the feasibility of implementing the Brazilian adaptation of the Irish intervention "iHELP Stroke: Improving Health and Lifestyle Programme", which aims to promote the adoption of healthy lifestyle behaviors post-stroke.

Methodology: This is a phase 1 interventional feasibility study, using a pre- and post-intervention design, to be conducted with ten individuals post-stroke, residing in Belo Horizonte, MG, Brazil. The intervention will consist of eight sessions: one educational session, one individual session, and six group sessions, held weekly. The outcomes of interest will include feasibility (recruitment, intervention, and measurement) and clinical outcomes (achievement of the main goal defined by the participants and the number/proportion of participants who meet this goal). Descriptive statistics will be used for analysis.

Conclusions: The results of this feasibility study will provide valuable insights for designing subsequent phases of a clinical trial.

DETAILED DESCRIPTION:
A non-probabilistic sample will be recruited from the community. Recruitment strategies include: referrals (e.g, phone numbers obtained from other research projects and university extension programs) and advertisements (e.g. physical folders distributed in public places and electronic pamphlets published on social media). All subjects will be informed about the study procedures and will provide written consent. The intervention and data collection will take place in a university laboratory setting. Two research assistants will enter the data into a statistical software package and verify any missing or apparently wrong values. Original paper forms will be kept in a secure place. Electronic files will be available only to the research team. All individuals will receive an identification code to ensure anonymity. A researcher, not involved in carrying out the intervention, will be responsible for carrying out the statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of subacute or chronic stroke;
* Age ≥ 18 years;
* Discharged from hospital and living in the community;
* Self-identified need to change at least one of the following lifestyle-related behaviors: physical inactivity, unhealthy diet, smoking, harmful alcohol use, or non-adherence to prescribed medication.

Exclusion Criteria:

* Positive screening test for possible cognitive alterations;
* Pain or other adverse health conditions that compromise the performance of the proposed intervention program, such as vestibular disorders, severe arthritis, or any other diagnosed disease of the nervous system;
* Presence of comprehensive and/or expressive aphasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Until the main outcome assessment period, which is 3 months.
  It will be determined by the ratio between the total number of eligible individuals (EI) and the total number of screened individuals (SI) (measure=EI/IS), and by the ratio between the total number of eligible individuals (EI) and the total number of recruited individuals (RI) (measure=EI/RI).
Feasibility of intervention (retention) | At baseline and post-intervention (week-8).
  It will be determined by the ratio between the total number of individuals who completed the proposed intervention program and the total number of individuals who started the proposed intervention program.
Feasibility of intervention (attendance) | At baseline and post-intervention (week-8).
  It will be determined by the ratio between the total number of sessions performed and the total number of sessions offered.
Feasibility of intervention (safety: incidence of treatment-emergent adverse events) | During the intervention (8 weeks).
  It will be determined by the number and reasons of adverse events (e.g. pain, falls, hospitalization, and death) identified during the period of intervention and follow-up of the individual.
Feasibility of intervention (perceived effectiveness) | At post-intervention (week-8).
  It will be determined by the following question: "Comparing how it was before you performed the intervention and now, do you consider your lifestyle to be healthier: strongly agree, partially agree, agree, neither agree nor disagree, disagree, partially disagree, strongly disagree."
Feasibility of measurement | At baseline and post-intervention (week-8).
  It will be determined by the percentage of clinical outcomes measured (ratio between the number of clinical outcomes measured and the number of clinical outcomes proposed to be measured).

SECONDARY OUTCOMES:
Achievement of the main goal defined by the participants | At baseline and post-intervention (week-8).
  Goal Attainment Scaling (GAS). The following scores will be identified: initial (or basal) T-score, final (or achieved) T-score, and T-score change (difference between the two measures). These scores will be calculated for all participants in order to identify the degree of achievement of the previously established main goal.
Number and proportion of participants who achieved their previously defined goals | At baseline and post-intervention (week-8).
  It is possible to categorize the final T-score based on the following classification: goal not achieved, when the T-score < 50; and goal achieved, when the T-score ≥ 50. Based on this classification, participants will be categorized according to the final (or achieved) T-score, in order to identify the number and proportion of individuals who met the previously defined main goal.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall P, Lawrence M, Kroll T, Blake C, Matthews J, Lennon O. Reducing risk behaviours after stroke: An overview of reviews interrogating primary study data using the Theoretical Domains Framework. PLoS One. 2024 Apr 26;19(4):e0302364. doi: 10.1371/journal.pone.0302364. eCollection 2024. PMID 38669261
- [Background] da Cruz Peniche P, Faria CDCM, Hall P, Lennon O. Effectiveness of behavior change and self-management theoretically-informed telehealth interventions for stroke secondary prevention: An overview of systematic reviews. J Telemed Telecare. 2025 Aug;31(7):961-990. doi: 10.1177/1357633X241238779. Epub 2024 Apr 16. PMID 38627913
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Moore G, Campbell M, Copeland L, Craig P, Movsisyan A, Hoddinott P, Littlecott H, O'Cathain A, Pfadenhauer L, Rehfuess E, Segrott J, Hawe P, Kee F, Couturiaux D, Hallingberg B, Evans R. Adapting interventions to new contexts-the ADAPT guidance. BMJ. 2021 Aug 3;374:n1679. doi: 10.1136/bmj.n1679. PMID 34344699